CLINICAL TRIAL: NCT01139203
Title: Prophylaxis of Hepatitis B Virus Recurrence After Liver Transplantation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Collaborators: Zhejiang University (Other)
Responsible Party: Shanghai First People's Hosptial
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: SH20100601
Record Dates: First submitted 2010-06-07; First posted 2010-06-08 (Estimated); Last update posted 2010-06-28 (Estimated); Status verified 2009-08

CONDITIONS: Liver Transplantation; Hepatitis B
Keywords: HBV recurrence; entecavir
MeSH Terms: conditions — Hepatitis B

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor

ARMS (3):
- lamivudine (Active Comparator)
  Interventions: Drug: lamivudine adefovir entecavir HBIG
- lamivudine and adefovir (Active Comparator)
  Interventions: Drug: lamivudine adefovir entecavir HBIG
- entecavir (Active Comparator)
  Interventions: Drug: lamivudine adefovir entecavir HBIG

INTERVENTIONS:
Drug: lamivudine adefovir entecavir HBIG — lamivudine 100mg orally daily adefovir 10mg orally daily entecavir 0.5mg orally daily HBIG 2000 unit intravenously during the anhepatic phase,and followed 800 unit intramuscularly daily until day 14,then 400 unit intramuscularly twice weekly

SUMMARY:
Entecavir demonstrated superior virologic and biochemical benefits over lamivudine and adefovir. The investigators evaluated the effect of entecavir combined Hepatitis B immune globulin (HBIG) with lamivudine or adefovir or both combined HBIG in Chinese liver transplantation patients with Hepatitis B Virus (HBV) related diseases.

ELIGIBILITY:
Inclusion Criteria:

1. patients into the transplant waiting list with HBV-related liver disease.
2. HBsAg-positive.
3. serum HBV-DNA negative.
4. no HCV, HDV and HIV co-infection.
5. without renal dysfunction.
6. No lamivudine, adefovir and entecavir drug allergy history.
7. no HBV-YMDD mutation for patients who have a long-term use of lamivudine.

Exclusion Criteria:

1. patients with HBV-related hepatocellular carcinoma beyond Milan criteria.
2. HBsAg-negative.
3. serum HBV-DNA positive.
4. HCV, HDV and HIV co-infection.
5. patients with severe renal dysfunction or failure.
6. lamivudine, adefovir and entecavir drug allergy history.
7. HBV-YMDD mutation for patients who have a long-term use of lamivudine.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2009-08; Primary Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
serological markers of HBV | every three month after liver transplantation
  Serological markers of HBV include HBsAg,HBsAb,HBeAg,HBeAb,HBcAb and HBV-DNA.

CONTACTS AND LOCATIONS:
Overall Officials: Zhi-Hai Peng, MD PHD, Study Chair — Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Locations (1):
- Shanghai First People's Hospital, Shanghai, China

REFERENCES:
- [Background] Patterson SJ, Angus PW. Post-liver transplant hepatitis B prophylaxis: the role of oral nucleos(t)ide analogues. Curr Opin Organ Transplant. 2009 Jun;14(3):225-30. doi: 10.1097/MOT.0b013e32832b1f32. PMID 19373086
- [Background] Angus PW, Patterson SJ. Liver transplantation for hepatitis B: what is the best hepatitis B immune globulin/antiviral regimen? Liver Transpl. 2008 Oct;14 Suppl 2:S15-22. doi: 10.1002/lt.21614. PMID 18825721
- [Background] Riediger C, Berberat PO, Sauer P, Gotthardt D, Weiss KH, Mehrabi A, Merle U, Stremmel W, Encke J. Prophylaxis and treatment of recurrent viral hepatitis after liver transplantation. Nephrol Dial Transplant. 2007 Sep;22 Suppl 8:viii37-viii46. doi: 10.1093/ndt/gfm655. PMID 17890261
- [Background] Carey I, Harrison PM. Monotherapy versus combination therapy for the treatment of chronic hepatitis B. Expert Opin Investig Drugs. 2009 Nov;18(11):1655-66. doi: 10.1517/13543780903241599. PMID 19852566